CLINICAL TRIAL: NCT05524233
Title: Transcranial Direct Current Stimulation (tDCS) For Improvement Of Cognitive Functioning, Brain Fog, And Working Memory
Brief Title: Transcranial Direct Current Stimulation (tDCS)
Acronym: tDCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Bijan Najafi, PhD, Professor of Surgery, Baylor College of Medicine, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 52200
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Results first posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Brain Fog
Keywords: Cognitive impairment; Brain fog; Transcranial stimulation
MeSH Terms: conditions — Mental Fatigue; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: All participants will be part of the intervention group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transcranial Direct Stimulation (Experimental): Subjects will receive an active electrical stimulation device (tDCS) to use up to 20 minutes daily for 4 weeks. To deliver tDCS subjects will place a strap around their forehead area.
  Interventions: Device: Active Transcranial Direct Stimulation

INTERVENTIONS:
Device: Active Transcranial Direct Stimulation — Subjects will receive a stimulation device to use up to 20 minutes daily for 4 weeks.

SUMMARY:
Cognitive impairment refers to when an individual struggles to learn, concentrate, remember, or make decisions. This can be due to underlying neurological diseases (i.e. Alzheimer's disease, dementia, etc.), caused by viral illness (i.e. brain fog experienced by COVID-19 survivors) or physical trauma (i.e. concussion). Recent reports indicate that two out of three Americans experience some amount of cognitive impairment in their lifetime.

There are a number of therapies that have been used to help address this condition. One of these is transcranial direct current stimulation (tDCS), which delivers sustained direct current to to the head area via electrodes. A number of studies have indicated that this form of therapy is safe and efficacious at inducing neuroplasticity and exciting neuronal activity. These factors can help improve aspects of cognitive functioning such as working memory, learning, and task performance.

The purpose of this pilot study is to examine the acceptability and proof of concept effectiveness of a wireless, transcranial direct current stimulation for people with cognitive impairments.

DETAILED DESCRIPTION:
Sample size (n=10) is convenient and designed to explore acceptability and feasibility. Participants who are enrolled will be provided a tDCS device to use for a period of four weeks. They will have two study visits, baseline (BL) and the 4th week visit (W4). During each visit participants will answer various questionnaires to assess patient-reported outcomes such as sleep quality, cognitive impairment, depression, anxiety, fatigue, and user acceptability.

The entire cohort will receive a transcranial direct stimulation (tDCS) device which uses LIFTiD Neurostimulation technology (RPW TECHNOLOGY, LLC, New York, USA). Participants will take the device home and daily, they will use the device for a maximum of 20 minutes to stimulate neuroplasticity. During the stimulation period they will be asked to perform a light activity such as reading, checking emails, etc. The participants will return to the McNair Campus for their final visit after 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adults (aged 18+) suffering from poor working memory, brain fog, or cognitive impairments (such as dementia, Alzheimer's, concussions, etc); ability to attend to the clinic for visits

Exclusion Criteria:

* Severe cognitive decline that reduces their ability to interact with the tDCS device; Major visual or hearing weakness reduces the ability to interact with tDCS device; Major foot problems such as active lower extremity wounds, major foot deformity (e.g., Charcot Foot), previous major amputations, and claudication; Demand-type cardiac pacemaker, implanted defibrillator, implanted metal plate in the brain or head, or other implanted electronic devices; Epilepsy, seizures, brain lesions, or severe heart disease; Sensitive skin or rash, broken skin, or open wounds; Pregnancy; and any conditions that may interfere with outcomes or increase the risk of the use tDCS based on the judgement of clinicians

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-09-29 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-04-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Transcranial Direct Stimulation
Started | 10
Completed | 5
Not Completed | 5
Not completed — Lost to Follow-up | 2
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Transcranial Direct Stimulation
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
MOCA Score [Mean (Standard Deviation); unit: units on a scale] — The Montreal Cognitive Assessment (MoCA) is a screening tool for mild cognitive impairment, assessing memory, attention, language, visuospatial skills, and executive functions. Scores range from 0 to 30, with 26 or above considered normal. Lower scores may indicate cognitive impairment: mild (19-25), moderate (10-18), and severe (below 10).
  units on a scale | 26.3 (3.92)

OUTCOME MEASURES:

1. Primary Outcome: Perceived Ease of Use After 4 Weeks of Daily tDCS Use (TAM Score)
Description: The perceived ease of use of tDCS will be assessed using a subscore of the Technology Acceptance Model (TAM) questionnaire.
  Participants will rate the device on a 5-point Likert scale (1 = Extremely Difficult, 5 = Extremely Easy) across seven questions. The total score will range from 7 (extremely difficult) to 35 (extremely easy), with higher scores indicating greater ease of use. Questions will assess: (1) ease of use, (2) sponge preparation, (3) attaching sponges, (4) starting/stopping therapy, (5) charging, (6) mobility while wearing the device, and (7) task completion during use.
  The TAM subscore will be calculated by summing individual scores, with median values reported as an overall measure of ease of use.
Time Frame: At 4 weeks
Population: The population includes the participants that completed the study.
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Transcranial Direct Stimulation
Number analyzed (Participants) | 5
units on a scale | 30.5 (4.8)

2. Primary Outcome: Perceived Usefulness After 4 Weeks of Daily tDCS Use (TAM Score)
Description: The perceived usefulness of tDCS was assessed using a subscore of the Technology Acceptance Model (TAM) questionnaire.
  Participants rated the usefulness of the device on a 5-point scale: 1 = Decreased Significantly, 2 = Decreased, 3 = Neutral, 4 = Increased, 5 = Increased Significantly. Six questions were used to assess overall perceived usefulness, focusing on benefits related to mental activity, energy levels, memory, attention, concentration, and alertness. The total score ranged from 6 (not at all useful) to 30 (highly useful), with higher values indicating greater perceived usefulness.
  The TAM subscore for perceived usefulness was calculated by summing the individual component scores and determining the median value across participants.
Time Frame: At 4 weeks
Population: The population includes the participants that completed the study.
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Transcranial Direct Stimulation
Number analyzed (Participants) | 5
units on a scale | 22.5 (4.5)

3. Primary Outcome: Attitude Towards Use After 4 Weeks of Daily tDCS Use (TAM Score)
Description: The attitude toward use of the tDCS device was assessed using a subscale of the Technology Acceptance Model (TAM) questionnaire.
  Participants will rate their attitude toward use on a 5-point Likert scale (1 = Extremely Difficult, 5 = Extremely Easy) based on two questions: (1) I would continue this therapy after completing the study, and (2) I would recommend this therapy to friends/family. The total score ranges from 2 (extremely difficult) to 10 (extremely easy), with higher scores reflecting a more positive attitude toward the device.
  The TAM subscore is calculated by summing individual component scores, with median values reported, providing an overall measure of perceived ease of use and intention to use.
Time Frame: At 4 weeks
Population: The population includes the participants that completed the study.
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Transcranial Direct Stimulation
Number analyzed (Participants) | 5
units on a scale | 9 (3.5)

4. Secondary Outcome: Change in Digit Memory Test Average Score at 4 Weeks Compared to Baseline
Description: A digit memory test assesses short-term and working memory by having participants recall sequences of numbers presented in either the same order (forward) or reverse order (backward). Scores are based on the longest sequence accurately recalled, with higher scores indicating better memory capacity. This test is commonly used in cognitive evaluations and research to monitor memory function and detect impairments. Percentage of changes in the total score were assessed at the 4-week mark compared to baseline. The range will be -100% to +100%. A score of zero indicates no change in memory performance, positive values reflect improvement, and negative values indicate a decline in memory performance.
  The average scores for all analyzed participants were reported.
Time Frame: Baseline - 4 weeks
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Transcranial Direct Stimulation
Number analyzed (Participants) | 5
Percent change | 2.5 (11.4)

5. Secondary Outcome: Change in Hopkins Verbal Learning Test Total Score at 4 Weeks Compared to Baseline
Description: The Hopkins Verbal Learning Test-Revised (HVLT-R) is a brief neuropsychological tool assessing verbal learning and memory. Participants recall 12 words across three trials (max score: 36) and a delayed recall trial (max score: 12), yielding a total score of 48, with higher scores indicating better memory.
  Percentage changes in cumulative scores from baseline to week 4 were evaluated, with averages reported across all participants who completed the study. Scores range from -100% to +100%, where positive values indicate improvement, zero denotes no change, and negative values reflect a decline.
Time Frame: Baseline - 4 weeks
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Transcranial Direct Stimulation
Number analyzed (Participants) | 5
Percent change | 45.8 (27.3)

6. Secondary Outcome: Changes in Trail Making Task (TMT) From Baseline
Description: The Trail Making Task (TMT) is a neuropsychological test used to assess attention, processing speed, and task-switching. It consists of two parts: Part A (connecting numbered circles sequentially) and Part B (alternating between numbers and letters). Performance is measured in seconds (completion time) and errors, with shorter times and fewer mistakes indicating better cognitive function. This study reported changes in TMT completion times at week 4 compared to baseline for both parts. Negative values indicate improvement (reduction in completion time compared to baseline) in cognitive function.
Time Frame: Baseline - 4 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Transcranial Direct Stimulation
Number analyzed (Participants) | 5
seconds
  Part A | -0.9 (11.5)
  Part B | -4.8 (15.3)

7. Other Pre Specified Outcome: Change in MoCA Score at 4 Weeks Compared to Baseline
Description: Cognitive status was assessed using the Montreal Cognitive Assessment (MoCA), which provides a score ranging from 0 to 30. Changes in scores from baseline to week 4 were reported, with positive values indicating improvement and negative values reflecting deterioration.
Time Frame: Baseline - 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transcranial Direct Stimulation
Number analyzed (Participants) | 5
score on a scale | -0.33 (1.63)

ADVERSE EVENTS:
Time Frame: up to 4 weeks post initiation of intervention
Description: The definition used will be the same as the clinicaltrials.gov definition.
Arm/Group | Transcranial Direct Stimulation
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 2/10
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transcranial Direct Stimulation (N=10)
Headches (General disorders) | 1 (1) — One participant experienced headaches during and after the initiation of electrical stimulation.
Pain (General disorders) | 1 (1) — One participant experienced skin pain during electrical stimulation.

LIMITATIONS AND CAVEATS:
Five participants (out of 10 baseline participants) were withdrawn for the following reasons: loss to follow-up (n=2), headache (n=1), skin irritation (n=1), and withdrawal of consent due to concerns about potential side effects (n=1). Consequently, only five participants completed the 4-week therapy and were included in the final analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-18): https://cdn.clinicaltrials.gov/large-docs/33/NCT05524233/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-27): https://cdn.clinicaltrials.gov/large-docs/33/NCT05524233/ICF_001.pdf